CLINICAL TRIAL: NCT04339075
Title: Registry to Investigate the Efficacy and Safety of VenaBlock VeIn SEaling System for VaRicose Veins in SingApore
Acronym: RIVIERA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2749
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Varicose Veins; Venous Reflux; Chronic Venous Insufficiency
Keywords: Endovenous Ablation
MeSH Terms: conditions — Varicose Veins | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Venablock: Patients that have undergone Venablock treatment
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires to access the quality of life (EQ5D, VCSS, CVVQ, CIVIQ, Patient satisfaction survey)

SUMMARY:
To assess the efficacy of the Venablock©Vein Sealing System (VBVS) for the treatment of lower extremity superficial truncal veins in a real-world clinical setting in a multi-racial Asian population in Singapore.

DETAILED DESCRIPTION:
The purpose of the Registry to Investigate the Efficacy and Safety of Venablock©Vein Sealing System for Varicose Veins in Singapore (RIVERIA), is to investigate the performance of cyanoacrylate glue closure (CAC) using this device, in which multiple incompetent superficial saphenous truncal veins (great saphenous (GSV), short saphenous vein (SSV), anterior accessory saphenous vein (AASV) will be treated at the same setting, and compression stockings will not be used post-operatively. The inclusion criteria for this study will be liberalized, and veins up to 12mm in diameter will be treated. As such,RIVIERA will be the first prospective trial conducted in Asia on a predominantly Asian cohort of patients to report on the performance of Venablock© for blocking incompetent truncal veins. This study specifically focuses on the initial technical outcomes, safety, anatomical occlusion, and patient experience after treatment with Venablock© with broader inclusion of patients than previous caucasian based trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 21 years old and ability to understand the requirements of the study and to provide informed consent
2. C2-C6 varicose veins/CVI (CEAP Class 1 patients will be excluded)
3. Symptomatic primary GSV,SSV or AASV incompetence, with reflux > 0.5 seconds on colour Duplex, including one or more of the following symptoms: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling
4. Patients who had GSV, SSV or AASV diameters of 3mm to 12mm in the standing position

Exclusion Criteria:

1. Current DVT or history of DVT
2. Pregnant patients
3. Arterial disease (ABPI<0.8)
4. Sepsis
5. Patient who are unwilling to participate
6. Inability or unwillingness to complete the time-point questionnaires
7. Adverse reaction to sclerosant or cyanoacrylate previously
8. Multiple drug allergies
9. Previous intervention with the VenaSeal cyanoacrylate glue closure system
10. Severely tortuous GSV, SSV or AASV
11. Life expectancy < 1 year
12. Active treatment for malignancy other than non-melanoma skin cancer
13. Current, regular use of systemic anticoagulation (e.g., warfarin, heparin)
14. Daily use of narcotic analgesia or NSAIDS to control pain associated with venous disease

Ages: 21 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will be undergoing Venablock© as a treatment for their varicose veins / chronic venous insufficiency
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Occlusion of treated vein post-procedure | Immediately post-op
Change in anatomy of treated vessel | 2 weeks, 3 months, 6 months, 12 months post-procedure
  Anatomical Success as measured at each timepoint using ultrasound to ensure occlusion of treated vessel. Recurrence or treatment failure will be defined as a re-opening of a segment > 5cm in length.

SECONDARY OUTCOMES:
Quality of Life Score using the EQ-5D questionnaire | 2 weeks, 3 months, 6 months, 12 months post-procedure
  EQ5D is used to assess quality of life based on Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety, rated at 5 levels: no problems, slight problems, moderate problems, severe problems, unable to perform activity. Inputs from this questionnaire is used to observe for changes in quality of life overtime. The higher the score, the better the quality of life is.
Quality of Life Score using the Chronic Venous Insufficiency Questionnaire (CIVIQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  CIVIQ is a questionnaire based on three dimensions - pain, physical and psychological, based on a scale from 1 to 5 (no trouble, slight, moderate, considerable, severe). Based on inputs, Global Index Score (GIS) will be tabulated, ranging for 0 to 100 - the higher the value, the poorer the quality of life.
Quality of Life score using the Aberdeen Varicose Vein Questionnaire (AVVQ) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  To measure health status of varicose veins patients based on symptoms and impact on daily activities. A total score ranging from 0 to 100 will be tabulated, with 100 being worst quality of life.
Clinical Change using Venous Clinical Severity Score (VCSS) | 2 weeks, 3 months, 6 months, 12 months post-procedure
  VCSS evaluates the severity of hallmarks of venous disease - 0 (none), 1 (mild), 2 (moderate), 3 (severe).
Pain Score | First 10 days post-procedure
  Using a numerical rating scale, which ranges from 0 (no pain) to 10 (severe pain)
Time taken to return to work and normal activities | Recorded 10 days post-procedure
Occlusion rates | 2 weeks, 3 months, 6 months, 12 months post-procedure
  Duplex ultrasound performed at specific timepoints to ensure that treated vein is occluded
Patient satisfaction with treatment: survey | 2 weeks, 3 months, 6 months, 12 months post-procedure
  A short survey to assess patient satisfaction and if there are any observed improvement in terms of appearance and symptoms post-procedure. Options range from highly unsatisfied to highly satisfied.
Cost effectiveness of the intervention | 12 months post-procedure
  to evaluate the cost involved with the procedure performed

CONTACTS AND LOCATIONS:
Overall Officials: Turn Yip Tang, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapre General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nesbitt C, Bedenis R, Bhattacharya V, Stansby G. Endovenous ablation (radiofrequency and laser) and foam sclerotherapy versus open surgery for great saphenous vein varices. Cochrane Database Syst Rev. 2014 Jul 30;(7):CD005624. doi: 10.1002/14651858.CD005624.pub3. PMID 25075589
- [Background] Siribumrungwong B, Noorit P, Wilasrusmee C, Attia J, Thakkinstian A. A systematic review and meta-analysis of randomised controlled trials comparing endovenous ablation and surgical intervention in patients with varicose vein. Eur J Vasc Endovasc Surg. 2012 Aug;44(2):214-23. doi: 10.1016/j.ejvs.2012.05.017. Epub 2012 Jun 15. PMID 22705163
- [Background] Darwood RJ, Theivacumar N, Dellagrammaticas D, Mavor AI, Gough MJ. Randomized clinical trial comparing endovenous laser ablation with surgery for the treatment of primary great saphenous varicose veins. Br J Surg. 2008 Mar;95(3):294-301. doi: 10.1002/bjs.6101. PMID 18278775
- [Background] Rasmussen LH, Lawaetz M, Bjoern L, Vennits B, Blemings A, Eklof B. Randomized clinical trial comparing endovenous laser ablation, radiofrequency ablation, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1079-87. doi: 10.1002/bjs.7555. PMID 21725957
- [Background] Marsden G, Perry M, Kelley K, Davies AH; Guideline Development Group. Diagnosis and management of varicose veins in the legs: summary of NICE guidance. BMJ. 2013 Jul 24;347:f4279. doi: 10.1136/bmj.f4279. No abstract available. PMID 23884969
- [Background] Shepherd AC, Gohel MS, Brown LC, Metcalfe MJ, Hamish M, Davies AH. Randomized clinical trial of VNUS ClosureFAST radiofrequency ablation versus laser for varicose veins. Br J Surg. 2010 Jun;97(6):810-8. doi: 10.1002/bjs.7091. PMID 20473992
- [Background] Shepherd AC, Gohel MS, Lim CS, Hamish M, Davies AH. Pain following 980-nm endovenous laser ablation and segmental radiofrequency ablation for varicose veins: a prospective observational study. Vasc Endovascular Surg. 2010 Apr;44(3):212-6. doi: 10.1177/1538574409359337. Epub 2010 Feb 11. PMID 20150227
- [Background] Rabe E, Otto J, Schliephake D, Pannier F. Efficacy and safety of great saphenous vein sclerotherapy using standardised polidocanol foam (ESAF): a randomised controlled multicentre clinical trial. Eur J Vasc Endovasc Surg. 2008 Feb;35(2):238-45. doi: 10.1016/j.ejvs.2007.09.006. Epub 2007 Nov 7. PMID 17988905
- [Background] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Background] Tang TY, Kam JW, Gaunt ME. ClariVein(R) - Early results from a large single-centre series of mechanochemical endovenous ablation for varicose veins. Phlebology. 2017 Feb;32(1):6-12. doi: 10.1177/0268355516630154. Epub 2016 Jul 9. PMID 26908638
- [Background] Vanlangenhove P, De Keukeleire K, Everaert K, Van Maele G, Defreyne L. Efficacy and safety of two different n-butyl-2-cyanoacrylates for the embolization of varicoceles: a prospective, randomized, blinded study. Cardiovasc Intervent Radiol. 2012 Jun;35(3):598-606. doi: 10.1007/s00270-011-0188-9. Epub 2011 Jun 3. PMID 21638147
- [Background] Brothers MF, Kaufmann JC, Fox AJ, Deveikis JP. n-Butyl 2-cyanoacrylate--substitute for IBCA in interventional neuroradiology: histopathologic and polymerization time studies. AJNR Am J Neuroradiol. 1989 Jul-Aug;10(4):777-86. PMID 2505505
- [Background] Ovali C, Sevin MB. Twelve-month efficacy and complications of cyanoacrylate embolization compared with radiofrequency ablation for incompetent great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2019 Mar;7(2):210-216. doi: 10.1016/j.jvsv.2018.10.019. Epub 2019 Jan 14. PMID 30655108
- [Background] Yavuz T, Acar AN, Aydin H, Ekingen E. A retrospective study of a new n-butyl-2-cyanoacrylate glue ablation catheter incorporated with application guiding light for the treatment of venous insufficiency: Twelve-month results. Vascular. 2018 Oct;26(5):547-555. doi: 10.1177/1708538118770548. Epub 2018 Apr 11. PMID 29642798
- [Background] Lee Q, Gibson K, Chan SL, Rathnaweera HP, Chong TT, Tang TY. A comparison between Caucasian and Asian superficial venous anatomy and reflux patterns - Implications for potential precision endovenous ablation therapy. Phlebology. 2020 Feb;35(1):39-45. doi: 10.1177/0268355519845984. Epub 2019 Apr 29. No abstract available. PMID 31032714